CLINICAL TRIAL: NCT02504411
Title: Outcomes of Disposable Distal Attachment Device (Endocuff and Transparent Plastic Cap) Assisted Colonoscopy Versus Standard Colonoscopy
Brief Title: Outcomes of Disposable Distal Attachment Device (Endocuff and Transparent Plastic Cap) Assisted Colonoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was not secured
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nirav C Thosani, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: HSC-MS-12-0587
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Device Assisted Colonoscopy (Experimental): Device assisted colonoscopy (DAC) is a technique of attaching disposable devices like "Endocuff" or "Transparent cap" at tip of colonoscope to improve mucosal visualization and stability.
  Interventions: Device: Device Assisted Colonoscopy
- Standard Colonoscopy (Active Comparator): Standard colonoscopy is the endoscopic examination of the large bowel and the distal part of the small bowel with a camera on a flexible tube passed through the anus.
  Interventions: Device: Standard Colonoscopy

INTERVENTIONS:
Device: Device Assisted Colonoscopy — This will be similar to the standard colonoscopy except the endocuff device will be used.
  Arms: Device Assisted Colonoscopy
Device: Standard Colonoscopy — No endocuff device will be used on the study participants undergoing standard colonoscopy.
  Arms: Standard Colonoscopy

SUMMARY:
The purpose of the study is to compare the efficacy of device assisted colonoscopy (DAC) with standard colonoscopy (SC) in detecting adenomas in a randomized fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing first screening colonoscopy
2. Patients undergoing subsequent surveillance colonoscopies with known history of prior colon polyps detected on prior screening colonoscopies.
3. Ability to provide informed consent.

Exclusion Criteria:

1. Previous surgical resection of any part of the colon
2. history of colon cancer
3. history of inflammatory bowel disease
4. use of antiplatelet agents or anti-coagulants that precluded removal of polyps
5. Poor general condition
6. History of polyposis syndrome or hereditary nonpolyposis colorectal cancer
7. Inability to give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) as determined by Colonoscopy | intraoperative
Complete adenoma resection rate (CARE) for adenoma > 10 mm in diameter as determined by Colonoscopy | intraoperative

SECONDARY OUTCOMES:
Cecal Intubation Rate (CIR) | intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Thosani, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States